CLINICAL TRIAL: NCT04649957
Title: Profiling the Determinants of Recovery to Establish Novel Rehabilitation Guidelines to Improve Clinically Relevant and Patient-reported Outcomes in the Post-COVID-19 Period
Brief Title: Profiling Recovery of Those Discharged Into the Community With COVID-19
Status: Completed | Type: Observational
Sponsor: University of Derby (Other)
Collaborators: Sheffield Hallam University (Other); University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mark Faghy, Senior Lecturer in Exercise Physiology, University of Derby
Other Study IDs: COVID-19-UoD&RDH20/21
Record Dates: First submitted 2020-12-01; First posted 2020-12-02 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Infections, Respiratory; Respiratory Physiology; Respiratory Muscle; Symptoms and General Pathology
Keywords: Respiratory; COVID-19; Recovery; Functional Status
MeSH Terms: conditions — Respiratory Tract Infections; Pathological Conditions, Signs and Symptoms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort Observation: Study investigators will identify eligible participants within 72 hours of expected discharge from hospital. Eligibility will be determined using the criteria outlined in section 5.1 which incorporates the Post-COVID-19 Functional Status (PCFS) Scale, a tool which has been developed and endorsed by the European Respiratory Society to measure functional status over time following COVID-19 infection. Patients graded 2, 3 or 4 on the PCFS will be eligible for participation. Eligible patients will be provided with a detailed explanation of the study including the provision of written information (PIS). Patients will be given time to consider participation in the research study before being approached again by the research team.
  If the patient expresses an interest in study participation the research team will invite participants to a baseline data collection session that will be held at the University of Derby (Kedleston Road campus) in the days following discharge.

SUMMARY:
Currently, there are few studies that have been established that consist of a variety of established and coherent approaches that sought to profile the determinants of recovery, nor used interrogative procedures to understand lasting physical impairment. In this context, measurements obtained from an assessment of cardio-respiratory responses to physiological stress could provide an important insight regarding the integrity of the pulmonary-vascular interface and characterisation of any impairment or abnormal cardio-respiratory function [4]. Indeed, current approaches are being developed to support patients using previous knowledge from other acute respiratory infections (e.g. Acute Respiratory Distress Syndrome; ARDS and Middle Eastern Respiratory Syndrome; MERS), approaches that do not consider the novel challenges presented by COVID-19. The knowledge obtained from the proposed research plan will inform the development of COVID-19 specific rehabilitation and clinical management guidelines which can be implemented globally to increase patient wellbeing, physical capacity, and functional status which will be directly related national and international health and wellbeing, economical and societal impacts.

DETAILED DESCRIPTION:
3.1 Screening and Eligibility Assessment Study investigators will identify eligible participants within 72 hours of expected discharge from hospital. Eligibility will be determined using the criteria outlined which incorporates the Post-COVID-19 Functional Status (PCFS) Scale, a tool which has been developed and endorsed by the European Respiratory Society to measure functional status over time following COVID-19 infection. Patients graded 2, 3 or 4 on the PCFS will be eligible for participation. Eligible patients will be provided with a detailed explanation of the study including the provision of written information (PIS). Patients will be given time to consider participation in the research study before being approached again by the research team.

If the patient expresses an interest in study participation the research team will invite participants to a baseline data collection session that will be held at the University of Derby in the days following discharge.

3.2 Assessments: Upon enrolment, admission clinical data and the results of investigations undertaken as part of the participants' usual care, before study enrolment will be collected, as outlined below. In the days following discharge (2 +/- 2 days) participants will complete a baseline assessments and measurements, outlined below and in the schedule of procedures.

At days 14, 42, 70, 98 (+/- 2 days) participants will conduct a consultation via telephone where all scales and questionnaires completed at baseline will be repeated (see the schedule of procedures outlined below). The total duration of these consultations' will be 15 minutes each time.

At Days 28, 56, 84, 112, 140 and 168 (+/- 2 days) participants will be attend a face to face appointment at the University of Derby's Human Performance Unit where physiological, biological, cognitive, and patient-reported outcome measures will be completed (see the schedule of procedures outlined below).

Where face to face or telephone consultations fall over a weekend (Saturday or Sunday) these will be arranged to occur on either the Friday before or Monday after, as convenient for the participant, but not more than 2 days away from the original date. The total duration of these research assessments will be 60 minutes per visit. All follow up appointments will be confirmed one week before the scheduled date via telephone/e-mail consultation. Acting as a reminder and to confirm the availability of the patient.

Schedule of Procedures

3.2.1 Baseline Clinical Data: Data collected will include demographics, the pre-admission symptoms, pre-admission therapy, pre-admission exercise tolerance and performance status (retrospective assessment by the patient and/or representative 6 weeks preceding admission) level of educational attainment, past-medical history, time and route of admission, and in-hospital routine physiological observations (including heart rate, blood pressure, oxygen saturation, respiratory rate and temperature). To ensure consistent recording of data across participants, we will collect the first set of physiological observations taken at / closest to 08.00 am on the morning of discharge.

3.2.2 Routine Clinical Investigations: The results of clinical investigations routinely performed during the participants' hospital admission, including those performed before study enrolment, will be collected including; blood parameters on admission to hospital full blood count (FBC), d-dimers, ferritin and Interleukin 6 (IL-6) Lactate dehydrogenase (LDH). If a radiological investigation was performed, the first investigation following admission will be recorded.

3.2.3 Post-COVID-19 Functional Status (PCFS) Scale The Post-COVID-19 Functional Status (PCFS) Scale will be assessed upon discharge from the hospital and during each face to face visit to monitor direct recovery and to assess functional sequelae. The PCFS will evaluate the ultimate consequences of COVID-19 on functional status and supplement other instruments that measure quality of life, tiredness, or dyspnoea in the acute phase. The PCFS covers the full spectrum of functional outcomes and focuses on both limitations in usual duties/activities and changes in lifestyle in six scale grades. Briefly grade 0 reflects the absence of any functional limitation, and the death of a patient is recorded in grade D. Upward of grade 1, symptoms, pain or anxiety are present to an increasing degree. This has no effect on activities for patients in grade 1, whereas a lower intensity of the activities is required for those in grade 2. Grade 3 accounts for inability to perform certain activities forcing patients to structurally modify these. Finally, grade 4 is reserved for those patients with severe functional limitations requiring assistance with activities of daily living (ADL).

3.2.3 Biomarkers: In-line with the outlined biomarkers in section 3.2.1, participants will have a serum sample taken for the measurement of inflammatory and metabolic biomarkers, including full blood count (to determine neutrophil leukocyte ratio (NLR) and the polymorph lymphocyte ratio (PLR), C-reactive protein (CRP), ferritin, d-dimers, ferritin and Interleukin 6 will be at discharge (Day 0). These samples are in addition to those collected during routine clinical care. Blood will be aliquoted, frozen, and stored for batch testing of biomarkers. These biomarkers have been selected because it has previously been demonstrated to correlate with a persistent reduction in quality of life scores. Participants will be asked to provide permission for the retention of these samples and consent for their use in future COVID-19 research studies.

3.2.4 Quality of Life: The EQ-5D-5L is routinely used in the assessment of the quality of life in respiratory research and is available in more than 130 languages (EQ-5D-5L, Appendix XX). It comprises five dimensions (previously 3): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.

3.2.5 Lung and Respiratory Muscle Function: Full lung function tests including FEV1 (forced expiratory volume at one second), FVC (forced vital capacity), PEFR (peak expiratory flow rate), flow-volume curves, MIP (maximal inspiratory pressure) and MEP (maximum expiratory pressure) will be measured at the hospital visits conducted at Day 0, all subsequent follow up appointments. These spirometry measurements will be conducted by a suitably qualified individual, proficient in the use of the specific equipment and according to published standards.

3.2.6 Symptom Profile: Symptom profile will be measured twice at the discharge assessment (Day 0), to capture a) retrospective assessment by the patient of their symptom status 6 weeks before admission (essentially their baseline symptoms before acute illness or admission), and b) their current symptom status at the point of discharge from hospital), and once at each subsequent weekly follow-up contact (either hospital visit or telephone consultation).

Fatigue is a common complaint in patients recovering from an acute respiratory infection and is not adequately captured in general quality of life or specific recovery questionnaires. Participants will complete 2 separate measures of fatigue at discharge (Day 0) and each subsequent follow-up contact; (A) the Fatigue Assessment Scale (FAS), a self-reported questionnaire validated to assess presence and severity of fatigue; and (B) MFI-20. A 20 item self-reported questionnaire assessing fatigue across five aspects.

The Medical Research Council (MRC) Dyspnoea Scale (MRC) is a measure to grade the effect of breathlessness on the person's daily activities. The MRC is simple to administer and is a short 1-5 stage scale (1 item) and allows the person to state the extent to which their breathlessness affects their mobility.

3.2.7 Cognition: The Montreal Cognitive Assessment (MoCA) will be conducted at discharge (Day 0) and again at Day 168. To reduce the impact of learning effect 2 distinct versions of the MoCA will be used as recommended by the developers, one at point of discharge, and repeat assessment at 168-day follow-up. To allow accurate interpretation, highest educational level/attainment will be recorded during the data collection phase of the study (before discharge).

3.2.8 Functional Status: Two different assessments of lower extremity functional capacity will be conducted at each visit these are (A) the 6-minute walk test (6MWT) and (B) the timed up and go test (TUG). The 6MWT is a standardised and widely used measure of functional status in individuals with chronic disease such as chronic obstructive pulmonary disease, cystic fibrosis, congestive cardiac failure, peripheral vascular disease, and elderly. It has been previously used to assess response to interventions and predict morbidity and mortality. Participants will be given a shortened practice attempt (1-2 minutes) at the beginning of each of their assessment visits. This will not be recorded but will be performed to allow familiarisation with the assessment and repeated at each visit for consistency.

The TUG is reliable and reproducible and has been validated as a predictor of frailty and risk of falls in elderly adults. The TUG has several advantages over other measures, mainly its reproducibility and shorter assessment time. Its use at predicting functional status following pneumonia has not been assessed previously.

Participants will also be asked to self-report their return to functional activity and employment at each contact with the research team (telephone consultations and follow-up visits.) Each participant will be asked at each contact with the research team if they have returned to perform their activities of daily living to the same level as 6 weeks before admission, and if they have returned to their occupation (if employed.) The patient-reported date of return to these activities will also be recorded.

3.2.10 Sleep Behaviour: Participants will complete the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-report measure to assess sleep quality over a 4 week in period, throughout the intervention. The measure consists of 19 individual items, with a 0-3 interval scale and creates 7 components that produce one global score. The PSQI is reliable and valid in the assessment of sleep problems.

3.2.11 Patient Experiences of COVID-19 Recovery Patient experiences of their recovery will be recorded via a free text weekly diary. Patients will be asked to provide free-text details about their experience throughout the week and to highlight any perceived changes in their symptom profile, recovery, and quality of life.

3.4 Description of Statistical Method: Statistical analysis will be supervised by Dr Emma Sharpe at the University of Derby and conducted using SPSS version 26. This study is a prospective observational cohort study, designed to identify suitable tools and measures across different domains for assessing patient recovery from COVID-19. Descriptive statistics will be calculated for all outcomes of interest. These will be presented as proportions and means with standard deviations or medians with interquartile ranges, depending on the distribution of data. Data will be collected at baseline and via face to face visits occurring every 28 days (days 28, 56, 84 and 112) which will be interspersed with telephone consultations, again occurring each 28 days (days 42, 70 and 98). Categorical data will be assessed using Chi-squared tests, whilst continuous outcome data will be analysed using Independent samples t-test or Mann-Whitney U test depending on the distribution. All qualitative components will be grouped collated upon study completion and analysed using Interpretative Phenomenological Analysis (IPA) in accordance with the methods proposed by Smith, Flowers and Larkin (2009).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged >18 years, including immunocompromised patients
* Admitted to hospital for treatment for mild/moderate COVID-19 (from NLR and PLR ratios and grade 2, 3 or grade 4 using PCFS Scale).
* Chest radiograph/CT scan consistent with COVID-19 infection.
* Able to understand verbal or written information in English

Exclusion Criteria:

* Below 18 years of age
* No confirmed diagnosis of COVID-19.
* Achieving a grade 0 or 1 on the PCFS.
* Not admitted to hospital/critical care for treatment of COVID-19.
* Reduced or lack of mental capacity
* Not able to understand verbal or written information in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study investigators will identify eligible participants within 72 hours of expected discharge from hospital. Eligibility will be determined using the criteria outlined in section 5.1 which incorporates the Post-COVID-19 Functional Status (PCFS) Scale, a tool which has been developed and endorsed by the European Respiratory Society to measure functional status over time following COVID-19 infection. Patients graded 2, 3 or 4 on the PCFS will be eligible for participation. Eligible patients will be provided with a detailed explanation of the study including the provision of written information (PIS). Patients will be given time to consider participation in the research study before being approached again by the research team.
  If the patient expresses an interest in study participation the research team will invite participants to a baseline data collection session that will be held at the University of Derby (Kedleston Road campus) in the days following discharge.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Post-COVID-19 Functional Status (PCFS) Scale | 16 weeks
  The PCFS offers the full spectrum of functional outcomes, and focuses on both limitations in usual duties/activities and changes in lifestyle in six scale grades.

SECONDARY OUTCOMES:
EQ-5D-5L | 16 weeks
  The EQ-5D-5L is routinely used in the assessment of the quality of life in respiratory research and is available in more than 130 languages (EQ-5D-5L). It comprises five dimensions (previously 3): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Faghy, PhD, Principal Investigator — University of Derby
Locations (1):
- University of Derby, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not part of the study teams plans.

REFERENCES:
- [Derived] Thomas C, Faghy MA, Owen R, Yates J, Ferraro F, Bewick T, Haggan K, Ashton REM. Lived experience of patients with Long COVID: a qualitative study in the UK. BMJ Open. 2023 Apr 26;13(4):e068481. doi: 10.1136/bmjopen-2022-068481. PMID 37185640